CLINICAL TRIAL: NCT04790968
Title: Combined PSMA PET/MRI for Detection of Lymph Node Metastases in High-risk Prostate Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Haukeland University Hospital (Other); University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REK 50719
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Prostatic Neoplasms; Neoplasm Metastasis
Keywords: Diagnostic imaging; Positron-emission tomography; Magnetic Resonance Imaging; Prostate-specific antigen; Lymph Nodes; PSMA; PET; Molecular imaging
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PSMA-PET/MRI and PET/CT for detection of lymph node metastases. (Experimental): Each patients will undergo an MRI-, PET/MRI- and PET/CT-examination (on the same day) prior to treatment.
  Patients in the radiotherapy cohort will additionally undergo an MRI examination after hormonal treatment, before radiotherapy.
  Interventions: Diagnostic Test: PSMA-PET; Diagnostic Test: PSMA-PET/MRI; Diagnostic Test: PSMA-PET/CT

INTERVENTIONS:
Diagnostic Test: PSMA-PET — Prostate specific membrane antigen positron emission tomography
Diagnostic Test: PSMA-PET/MRI — Prostate specific membrane antigen positron emission tomography combined with magnetic resonance imaging
Diagnostic Test: PSMA-PET/CT — Prostate specific membrane antigen positron emission tomography combined with computed tomography imaging

SUMMARY:
For high-risk prostate cancer patients, detection of lymph node metastases is crucial to ensure optimal treatment.

Standard treatment for these patients is radiotherapy or surgery. The surgery involves resection of the prostate and the pelvic lymph nodes. Currently, the most reliable method to confirm lymph node metastases is by histologic examination of the resected lymph nodes. Ideally, one should be able to detect lymph node metastases prior to treatment. Then, the treatment could be better adjusted to each patient.

Imaging methods such as prostate specific membrane antigen positron emission tomography (PSMA-PET) can possibly aid the detection of lymph node metastases. In this study, the investigators want to test whether PSMA-PET or a combination of PSMA-PET and MRI (magnetic resonance imaging) can improve staging of lymph nodes before treatment.

DETAILED DESCRIPTION:
High-risk prostate cancer patients have a high probability for lymph node metastases in the pelvic region. The lymph node status is an important prognostic factor in determining the risk of later relapses and a factor in treatment planning. Lymph node metastases outside the pelvis usually signify systemic treatment not amendable for curative treatment.

High-risk prostate cancer patients are treated by radiotherapy or surgical resection of the prostate and the pelvic lymph nodes. Currently, the most reliable method for confirming lymph node metastases is by bilateral pelvic lymph node dissection during surgical treatment, and subsequent histologic examination. However, todays state-of-the art methods for the detection of lymph node metastases prior to treatment are clearly inadequate. Detection of lymph node metastases is crucial for determining whether the patient (i) is a candidate for localized treatment and, if so, (ii) optimizing the extent of the lymph node dissection / radiation field for localized treatment. Non-standard imaging methods such as prostate specific membrane antigen (PSMA)-PET-imaging have been shown to be able to aid in the detection of lymph node metastases. The purpose of this study is to test whether PSMA-PET or a combination of PSMA-PET and MRI can improve the sensitivity and specificity for pre-treatment lymph node staging in order to reduce both over- and undertreatment of high-risk prostate cancer patients.

In this multi-centre study, at least 80 patients with high-grade prostate cancer (according to NCNN Guidelines, v 2.2022) will be examined with PSMA PET/MRI and PET/CT. Study recruitment will continue until 60 patients have received radial prostatectomy with extended pelvic lymph node dissection (ePLND) (surgery cohort) and 20 patients have been treated with radiotherapy to the prostate and pelvic lymph nodes (radiotherapy cohort). After the PET examinations, all patients will receive standard treatment and follow-up, which is determined by national guidelines and the patient's treating urologist and/or oncologist. Imaging data will be analyzed by radiologists and nuclear medicine physicians in collaboration. The imaging findings in the surgery cohort will be compared to the histology outcome after ePLND to assess the sensitivity and specificity for detection of lymph node involvement with PSMA PET/MRI. The data from the radiotherapy cohort will be used to assess the feasibility of PSMA PET/MRI-based radiotherapy planning. Advanced image processing and analysis methodology including the use of artificial intelligence will also be applied.

ELIGIBILITY:
Inclusion criteria (surgery cohort):

* High risk localized/locally advanced prostate cancer patients who are candidates for radical prostatectomy plus bilateral extended PLND; ISUP Gleason grade group ≥ 4

Inclusion criteria (radiotherapy cohort):

* High-risk localized/locally advanced prostate cancer patients scheduled for radiation treatment of the prostate and pelvic lymph nodes; ISUP Gleason grade group ≥ 4

Exclusion criteria (surgery and radiotherapy cohort):

* Prior history of any other cancer the last 5 years excluding basal cell carcinoma
* Proven metastases in bones or other distant metastases
* General contra-indications for MRI (pacemaker, aneurysm clips, any form of metal in the body, severe claustrophobia)
* Serious concomitant systemic disorders that in the opinion of the investigator would compromise the patient's ability to complete the study or interfere with the evaluation of the efficacy and safety of the study objectives
* Metal implants in the pelvic region which will deteriorate PET/MR/CT image quality.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of PSMA PET and combined PSMA PET/MRI | 1 month
  To compare the diagnostic accuracy of PSMA PET and combined PSMA PET/MRI to that of the current standard multiparametric MRI, using histopathology as the gold standard.

SECONDARY OUTCOMES:
Sensitivity and specificity of PSMA PET/MRI | 1 month
  To evaluate the sensitivity and specificity of PSMA PET/MRI to detect positive lymph nodes in high-risk prostate cancer patients in a prospective, multicenter study.
Performance of PSMA PET/MRI versus PET/CT | 1 month
  Compare the performance of PET/MRI to PET/CT for detection of lymph node metastases

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Risa, Prof, Study Director — Norwegian University of Science and Technology, NTNU; Morten Troøyen, MD, Study Director — St. Olavs Hospital
Locations (3):
- Norway (3):
  - Haukeland University Hospital, Bergen
  - University Hosptial of North Norway, Tromsø
  - St Olavs Hospital, Trondheim University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Undecided